CLINICAL TRIAL: NCT03655691
Title: Clinical Trial to Evaluate ET-01 in Subjects With Lateral Canthal Lines
Brief Title: ET-01 in Subjects With Lateral Canthal Lines, LCL-207
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eirion Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ET-01-LCL-207
Record Dates: First submitted 2018-08-30; First posted 2018-08-31 (Actual); Results first posted 2022-02-18 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Lateral Canthal Lines; Crow's Feet
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: parallel dose groups
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: different doses are packaged in identical containers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Vehicle (Placebo Comparator): Vehicle / Placebo formulation
  Interventions: Biological: Vehicle
- Dose 1 (Experimental): lower dose of ET-01
  Interventions: Biological: botulinum toxin, Type A
- Dose 2 (Experimental): higher dose of ET-01
  Interventions: Biological: botulinum toxin, Type A

INTERVENTIONS:
Biological: Vehicle — Vehicle Formulation
  Arms: Vehicle
Biological: botulinum toxin, Type A — botulinum toxin, Type A, lower Dose 1, administered once, topically, at Baseline
  Other Names: ET-01
  Arms: Dose 1
Biological: botulinum toxin, Type A — botulinum toxin, Type A, higher Dose 2, administered once, topically, at Baseline
  Other Names: ET-01
  Arms: Dose 2

SUMMARY:
This study tests an investigational drug formulation called ET-01, botulinum toxin, Type A, topical, in lateral canthal lines (LCL).

DETAILED DESCRIPTION:
This product is being tested for its ability to reduce lateral canthal lines, also known as Crow's Feet.

ELIGIBILITY:
Inclusion Criteria:

* 25 - 65 years of age
* minimal to moderate Crow's Feet wrinkles at rest
* moderate to severe Crow's Feet wrinkles on contraction
* willingness to refrain from any product affecting skin remodeling
* female subjects must be not pregnant and non-lactating

Exclusion Criteria:

* history of adverse reactions to any prior botulinum toxin treatments
* history of vaccination or non-response to any prior botulinum toxin treatments
* botulinum toxin treatment in the prior 6 months
* present or history of neuromuscular disease, eyelid ptosis, muscle weakness, paralysis, or "dry eye"
* history of peri-ocular surgery, brow lift or related procedures
* procedures affecting the lateral canthal region in the prior 12 months
* application of topical prescription medication to the treatment area
* female subjects who are pregnant or are nursing a child

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2018-11-09 (Actual); Study Completion 2019-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Theobald, MD, PhD, Study Director — Eirion Therapeutics
Locations (6):
- United States (6):
  - Baumann Cosmetic & Research Institute, Miami, Florida
  - Radiant Research, Inc., Pinellas Park, Florida
  - Research Institute of the Southeast, LLC, West Palm Beach, Florida
  - Dermatology NOLA Inc., Metairie, Louisiana
  - Westlake Dermatology Clinical Research Center, Austin, Texas
  - Virginia Clinical Research, Inc., Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from six medical centers between August and October 2018.
Pre-assignment Details: A total of N=104 subjects were screened; N=80 were found eligible; N=1 subject withdrew consent prior to treatment assignment; N=79 were randomized.
Groups:
- Vehicle: Vehicle / Placebo formulation
  Vehicle: Vehicle Formulation, administered once, topically, at Baseline
Period: Overall Study
Arm/Group | Vehicle | Dose 1 | Dose 2
Started | 26 | 26 | 27
Completed | 24 | 23 | 24
Not Completed | 2 | 3 | 3
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 1 | 2
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dose 2: higher dose of ET-01
  botulinum toxin, Type A: botulinum toxin, Type A, Dose 2, administered once, topically, at Baseline
- Total: Total of all reporting groups
Arm/Group | Vehicle | Dose 1 | Dose 2 | Total
Number analyzed (Participants) | 26 | 26 | 27 | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 25 | 26 | 26 | 77
  >=65 years | 1 | 0 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (9.0) | 51.3 (8.2) | 51.4 (7.3) | 50.6 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 24 | 21 | 65
  Male | 6 | 2 | 6 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 2 | 3
  White | 22 | 24 | 23 | 69
  More than one race | 3 | 2 | 0 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 26 | 26 | 27 | 79
IGA-C [Mean (Standard Deviation); unit: units on a scale] — Investigator Global Assessment on Contraction using the ordinal Crow's Feet Wrinkle Scale where severity is scored between 0=absent and 4=severe.
  units on a scale | 3.7 (0.4) | 3.6 (0.5) | 3.6 (0.5) | 3.6 (0.5)
SSA-C [Mean (Standard Deviation); unit: units on a scale] — Subject Self-Assessment on Contraction using the ordinal Crow's Feet Wrinkle Scale where severity is scored between 0=absent and 4=severe.
  units on a scale | 3.5 (0.5) | 3.8 (0.4) | 3.6 (0.5) | 3.6 (0.5)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Response Defined as Change in IGA-C (Investigators Global Assessment) Score by at Least 2 Ordinals From Baseline to Week 4
Description: Investigators Global Assessment of the Crow's Feet Wrinkle Scale where severity is scored between 0-4 (0=absent; 4=severe). Response is defined as change by at least two ordinals from Baseline to Week 4.
Time Frame: Week 4
Population: Intent-To-Treat (ITT) population defined as all treated subjects who had at least one post-baseline visit. No imputation was performed when only incomplete data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle | Dose 1 | Dose 2
Number analyzed (Participants) | 24 | 26 | 26
Participants | 4 | 1 | 3

2. Secondary Outcome: Total Number of Observations With a Response Defined as IGA-C Score ≤ 2 at Any Time Between Week 2 and Week 18
Description: Total number of observations with a Score of ≤ 2 on the Investigators Global Assessment on Contraction, IGA-C, using the Crow's Feet Wrinkle Scale, where severity is scored between 0-4 (0=absent; 4=severe). To count, a "responder" is defined as Score ≤ 2. The observation period ranges from the earliest expected onset of action at Week 2 to the likely offset of action by Week 18.
Time Frame: Week 2, 4, 8,12, and 18
Population: as for outcome 1
Measure: Count of Units; unit: Observations
Units Other Than Participants: Observations
Arm/Group | Vehicle | Dose 1 | Dose 2
Number analyzed (Participants) | 24 | 26 | 26
Number analyzed (Observations) | 146 | 151 | 152
Observations | 33 | 18 | 44

3. Secondary Outcome: Total Number of Observations With a Response Defined as SSA-C Score ≤ 2 at Any Time Between Week 2 and Week 18
Description: Total number of observations with a Score of ≤ 2 on the Subjects Self-Assessment on Contraction, SSA-C, using the Crow's Feet Wrinkle Scale, where severity is scored between 0-4 (0=absent; 4=severe). To count, a "responder" is defined as Score ≤ 2. The observation period ranges from the earliest expected onset of action at Week 2 to the likely offset of action by Week 18.
Time Frame: Week 2, 4, 8,12, and 18
Population: as for outcome 1
Measure: Count of Units; unit: Observations
Units Other Than Participants: Observations
Arm/Group | Vehicle | Dose 1 | Dose 2
Number analyzed (Participants) | 24 | 26 | 26
Number analyzed (Observations) | 146 | 151 | 152
Observations | 30 | 8 | 17

ADVERSE EVENTS:
Time Frame: 26 Weeks
Groups:
- Dose 1: lower dose of ET-01
  botulinum toxin, Type A: botulinum toxin, Type A, Dose 1
- Dose 2: higher dose of ET-01
  botulinum toxin, Type A: botulinum toxin, Type A, Dose 2
Arm/Group | Vehicle | Dose 1 | Dose 2
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26 | 1/27
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26 | 3/27
Other Adverse Events (participants affected / at risk) | 4/26 | 3/26 | 2/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle (N=26) | Dose 1 (N=26) | Dose 2 (N=27)
Accidental death (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Death by gunshot wound.
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Depression (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — worsening of pre-existing condition.
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle (N=26) | Dose 1 (N=26) | Dose 2 (N=27)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Large intestine benign neoplasm (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Study Results are considered Confidential Information that may not be published or disclosed without Sponsor's written consent for a period of five (5) years after completion of the Study.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-06): https://cdn.clinicaltrials.gov/large-docs/91/NCT03655691/Prot_SAP_000.pdf